CLINICAL TRIAL: NCT04830878
Title: A Phase I, Multicenter, Uncontrolled, Open Label Study Assessing the Efficacy and Safety of a Combination of Systemic and Intravitreal Injections of Methotrexate for the Prevention and Treatment of Proliferative Vitreoretinopathy in Pediatric Patients With RheGmatogenous Retinal DetacHmenT (the SIGHT Study)
Brief Title: Methotrexate For The Prevention and Treatment of Proliferative Vitreoretinopathy in Pediatric Patients
Acronym: SIGHT
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB-59989
Record Dates: First submitted 2021-03-31; First posted 2021-04-05 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Proliferative Vitreoretinopathy
MeSH Terms: conditions — Vitreoretinopathy, Proliferative | interventions — Methotrexate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Methotrexate treatment
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Methotrexate — Systemic and intraoperative intravitreal injection of methotrexate

SUMMARY:
Rhegmatogenous retinal detachment (RRD) is a sight-threatening condition. Children with RRD usually present late with clinical features of longstanding RRD, specifically a serious condition named: proliferative vitreoretinopathy (PVR). Therefore, children with RRD often have poorer outcomes. The objective of this study is to investigate the efficacy and safety of methotrexate in the treatment and prevention of PVR. Methotrexate is a medication that has been used to treat inflammatory conditions in children and adults for a long time and it has been recently used to treat PVR in adults.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to get informed consent from a parent or a legal guardian of the child and attend all study visits.
2. Males or females 18 years old or younger.
3. Subject is undergoing vitrectomy for either i. initial retinal detachment with or without PVR ii. recurrent retinal detachment due to grade A or higher of proliferative vitreoretinopathy.
4. Female subjects of childbearing potential must not be pregnant or breast-feeding, must have a negative serum pregnancy test at screening, and must be willing to undergo pregnancy tests throughout the study.
5. Female subjects of childbearing potential and male subjects able to father children must (a) abstain from intercourse throughout the course of the study or (b) agree to practice acceptable methods of contraception throughout the course of the study (i.e., intrauterine device, oral contraceptives, barrier method, or other contraception deemed adequate by the investigator).

Exclusion Criteria:

1. Ocular or periocular infection in either eye including (but not limited to):

   1. History of herpetic infection in the study eye(s) or adnexa.
   2. Presence of known active or inactive toxoplasmosis or toxoplasmosis scar in either eye.
   3. History of cytomegalovirus infection or clinical evidence of active cytomegalovirus infection at screening and/or Day 1.
2. Pupillary dilation inadequate for quality stereoscopic fundus photography in the study eye(s).
3. Media opacity that would limit clinical visualization in the study eye(s) and, in the opinion of the investigator, could not be repaired or improved during the RD surgery.
4. Other planned eye surgery during the course of the trial
5. Corneal opacity in the study eye(s) that would preclude reliable assessment of the posterior segment.
6. Uncontrolled glaucoma in the study eye(s), evidenced by an intraocular pressure (IOP) > 21 mmHg while on maximum medical therapy, or chronic hypotony (unmeasurable eye pressure).
7. Subjects should not be currently undergoing treatment with one of the following at the time of RD diagnosis: systemic steroids, methotrexate, azathioprine, or mycophenolate mofetil (or an equivalent drug, e.g., mycophenolic acid) or other immunomodulatory therapies.
8. Malignancy in remission for less than 5 years prior to study participation.
9. Allergy or hypersensitivity to investigational product or other study related procedures/medications.
10. Any recent systemic infection (excluding common cold) within 30 days of Day 1.
11. Known to be immunocompromised.
12. History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease condition that contraindicates the use of an investigational drug, might affect the interpretation of the results of the study, or renders the subject at high risk for treatment complications.
13. Any uncontrolled systemic disease, except stable syndromic conditions.
14. Females who are pregnant or lactating and females of child-bearing potential who are not using adequate contraceptive precautions (i.e., intrauterine device, oral contraceptives, barrier method, or other contraception deemed adequate by the investigator).
15. Participation in other investigational drug (oral or topical therapy) or device clinical trials within 30 days prior to Day 1 and/or participation in other investigational drug (intravitreal injection therapy) within 3 months or 5 half-lives (whichever is longer) prior to Day 1 or planning to participate in other investigational drug or device clinical trials during a time which would overlap with the duration of the study. This includes both ocular and non-ocular clinical trials. Exposure to investigational biologics should be discussed with the investigators.
16. In addition, the investigator may declare a subject ineligible for any sound reason.
17. Chest X-ray within 3 months prior to initiation of systemic MTX that shows active pulmonary diseases of any etiology.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Recurrence of Retinal Detachment | 6 months
  Number of Participants with Recurrent Retinal Detachment

CONTACTS AND LOCATIONS:
Overall Officials: Edward Wood, MD, Principal Investigator — Stanford University; Quan Dong Nguyen, MD, MSc, Principal Investigator — Stanford University; Ahmad Al-Moujahed, MD, PhD, MPH, Principal Investigator — Stanford University; Hashem Ghoraba, MD, Principal Investigator — Stanford University; Darius Moshfeghi, MD, Principal Investigator — Stanford University
Locations (1):
- Byers Eye Institute at Stanford University and Lucille Packard Children Hospital, Palo Alto, California, United States